CLINICAL TRIAL: NCT05296681
Title: A Randomized Trial of Microbiotic Product (NBT-NM108) to Promote Microbiome Health and Improve Chemotherapy Delivery
Brief Title: Microbiotic Product to Promote Microbiome Health and Improve Chemotherapy Delivery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Howard S. Hochster, MD (Other)
Responsible Party: Sponsor-Investigator, Howard S. Hochster, MD, Associate Director for Clinical Research and Director, GI Oncology, Rutgers Cancer Institute, Director of Oncology Research, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 072201; Pro2022000222 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colon Carcinoma; Stage IV Colon Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8
Keywords: chemotherapy-induced diarrhea
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive NBT-NM108 or no microbiome support in a 2:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NM108 Drinks (Experimental): NBT-NM108 Drinks four times daily before meals and 2 hours after dinner for 56 days.
  Beginning 5 days before starting chemotherapy, patients receive NBT-NM108 PO QID for 56 days. Patients receive irinotecan-based chemotherapy per standard of care.
  Interventions: Drug: NBT-NM108
- No Microbiome Support (No Intervention): No microbiome
  Patients receive irinotecan-based chemotherapy per standard of care.

INTERVENTIONS:
Drug: NBT-NM108 — Patients receive irinotecan-based chemotherapy per standard of care.
  Arms: NM108 Drinks

SUMMARY:
This phase II trial tests whether NBT-NM108 works in reducing chemotherapy-induced diarrhea in patients with colon cancer that has spread to other places in the body (metastatic). Irinotecan is one of the most used medicine for colon cancer, but it leads to diarrhea in most patients receiving it and among some of them, severe diarrhea can occur. NBT-NM108 is a high dietary fiber formula that is developed based on research findings that have shown that high fiber diets can help maintain healthy bacteria in the gut and improve gut function. Giving NBT-NM108 to patients with colon cancer receiving chemotherapy may help relieve or lessen diarrhea symptoms and lead to improved tolerance of the chemotherapy drug, irinotecan.

DETAILED DESCRIPTION:
PRIMARY ENDPOINT:

Dose Intensity of Irinotecan administered (mg/m2/week)

SECONDARY ENDPOINTS:

1. Reduction in % Patients Needing Dose Modification for Diarrhea
2. Toxicity Grade of diarrhea
3. Response Rate
4. Time to Progression-free survival

EXPLORATORY ENDPOINTS:

1. 16S rRNA gene sequencing to reveal changes of the gut microbiota including institution of foundation guilds and restoration of healthy microbiome
2. Short chain fatty acids analysis (promotion of acetic and butyric acid production)
3. Markers for gut inflammation such as fecal lipocalin 2
4. Gut barrier function test to see if the restoration of healthier gut microbiota would improve gut barrier function.

ELIGIBILITY:
Inclusion Criteria

* Biopsy proven and metastatic colon cancer
* Candidate for Second-line or later line therapy with irinotecan-based chemotherapy regimen with starting dose of irinotecan at 180 mg/m2 q2w.

Participants who have had prior irinotecan will be eligible if they are off irinotecan for at least three months and stools have returned to baseline consistency.

* Performance Status (PS) 0-1
* Lab values as acceptable for trials: Absolute Neutrophil Count( ANC) >1500/uL; Creatinine < 1.5 x Upper Limit of Normal (ULN); Transaminases < 5x ULN; Bilirubin < 1.5 x ULN; Albumin > 3.0 g/dL
* No known UGTA1A* genotype

Exclusion Criteria

* Grade two diarrhea or greater (4-6 movements per day over baseline)
* Inability to take oral supplements
* Current antibiotic therapy
* Baseline grade 3-4 diarrhea Participants with grade two diarrhea should undergo stool evaluation with stool test for bacteria (Salmonella, Shigella, Campylobacter, Yersinia Mycobacterium), bacterial toxin (Clostridium difficile), ova and parasites (Giardia, Entamoeba, Isospora, Cyclospora, Cryptosporidium, Microsporidium), or viruses (Cytomegalovirus), associated with an ongoing active infection and diarrhea. They will be eligible if this evaluation shows no infection.
* History of the following infections and/or disease which could lead to diarrhea:
* History of prior positive gastrointestinal biopsy, gastrointestinal culture, or stool test for bacteria (Salmonella, Shigella, Campylobacter, Yersinia, Mycobacterium), bacterial toxin (Clostridium difficile), ova and parasites (Giardia, Entamoeba, Isospora, Cyclospora, Cryptosporidium, Microsporidium), or viruses (Cytomegalovirus), associated with an ongoing active infection and diarrhea unless fully treated with at least three months normal stool.
* History of ulcerative colitis, Crohn's disease, celiac sprue (gluten-enteropathy), chronic pancreatitis, malabsorption, or any other gastrointestinal disease associated with diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants with treatment-related Adverse Events as Assessed by Cancer Therapy Evaluation Program Common Toxicity Criteria (CTCAE) Version 5.0 for toxicity and Adverse Event reporting | Eight weeks
  The number of participants with treatment-related Adverse Events as Assessed by Cancer Therapy Evaluation Program Common Toxicity Criteria (CTCAE) Version 5.0 for toxicity and Adverse Event reporting. Dose reduction should occur for CTCAE grade 3 or higher toxicity given maximum antidiarrheal support with Imodium and/or Lomotil.
Tumor Response by RECIST v1.1 Criteria | Imaging for response assessment will be obtained before the initiation of conditioning (no more than 4 weeks prior to apheresis) and at the 6-week follow up time point
  Response and progression will be evaluated in this study using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used for tumor measurements

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Hochster, MD, Principal Investigator — Rutgers University
Locations (10):
- United States (10):
  - Robert Wood Johnson University Hospital, Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Lakewood, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Cancer Center, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson University Hospital, Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No